CLINICAL TRIAL: NCT06010303
Title: A Phase 2, Randomized, Active-Controlled, Open-Label Study to Evaluate the Efficacy and Safety of LBL-007 in Combination With Tislelizumab Plus Chemotherapy as First-Line Treatment in Patients With Unresectable Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study to Evaluate LBL-007 in Combination With Tislelizumab Plus Chemotherapy in Participants With Unresectable Locally Advanced or Metastatic Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-LBL-007-202; CTR20233227 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Cancer; Esophageal Squamous Cell Carcinoma; Esophageal Squamous Cell Carcinoma by AJCC V8 Stage
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LBL-007 (Experimental): LBL-007 in combination with tislelizumab plus chemotherapy doublet.
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Chemotherapy Doublet
- Tislelizumab and Chemotherapy (Active Comparator): Tislelizumab plus chemotherapy doublet.
  Interventions: Drug: Tislelizumab; Drug: Chemotherapy Doublet

INTERVENTIONS:
Drug: LBL-007 — LBL-007 will be administered at a standard dose intravenously.
  Other Names: Alcestobart
  Arms: LBL-007
Drug: Tislelizumab — Tislelizumab will be administered at a standard dose intravenously.
  Other Names: BGB-A317
Drug: Chemotherapy Doublet — Doublet 1: cisplatin + 5-fluorouracil Doublet 2: cisplatin + paclitaxel
  Choice of chemotherapy doublet will be determined by the investigator and will be administered at standard doses intravenously.

SUMMARY:
This is a randomized, open-label study to compare how well LBL-007 works in combination with tislelizumab and chemotherapy versus tislelizumab and chemotherapy when given as the first-line treatment in participants with inoperable locally advanced or metastatic esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and can agree to comply with the study requirements.
* Participants with metastatic ESCC or unresectable, locally advanced ESCC.
* Histologically confirmed diagnosis of ESCC.
* Can provide a tumor sample.
* At least 1 measurable lesion as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.

Exclusion Criteria:

* Prior treatment for advanced or metastatic ESCC within the past 6 months
* Locally advanced ESCC that is either resectable or potentially curable with definitive chemoradiation treatment per local investigator
* Palliative radiation treatment for ESCC within the past 4 weeks
* Participants with an esophageal/bronchial or esophageal/aorta fistula
* Prior treatment with programmed cell death protein-1 (PD-1) or other immune-oncological drugs

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 10 months
  Percentage of participants whose best overall response (BOR) is complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 18 months
  Time from the date of randomization to the date of first documentation of disease progression assessed by the investigator per RECIST v1.1 or death, whichever occurs first.
Duration of Response (DOR) | Approximately 18 months
  Time from the first determination of an overall response until the first documentation of progression assessed by the investigator per RECIST v1.1 or death, whichever occurs first.
Disease Control Rate (DCR) | Approximately 18 months
  Percentage of participants whose BOR is CR, PR, and stable disease as assessed by the investigator per RECIST v1.1.
Number of Participants with Adverse Events (AEs) | Approximately 18 months
  Number of participants with AEs, including findings from physical examinations, electrocardiograms, and laboratory assessments according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (38):
- China (24):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital Branch North, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, Seoul, Seoul Teugbyeolsi
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (4):
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Hrh Princess Maha Chakri Sirindhorn Medical Center (Srinakharinwirot University), Ongkharak
  - Phramongkutklao Hospital, Ratchathewi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/